CLINICAL TRIAL: NCT04959812
Title: Analgesics in the Pre-hospital Setting: Implications on Hemorrhage Tolerance - Sufentanil
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU-2021-0579
Record Dates: First submitted 2021-06-29; First posted 2021-07-13 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sufentanil (Experimental): Sufentanil (30 microgram tablet) will be administered via a sublingual pill
  Interventions: Drug: Sufentanil
- Placebo (Placebo Comparator): Placebo will be administered via a sublingual pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sufentanil — Subjects will receive Sufentanil while the effects of this drug on tolerance to a hemorrhagic insult will be assessed.
  Arms: Sufentanil
Other: Placebo — Subjects will receive a placebo pill while the effects of this placebo on tolerance to a hemorrhagic insult will be assessed.
  Arms: Placebo

SUMMARY:
This study will examine how sufentanil (a commonly used pain medication) will alter responses to simulated blood loss in humans. To simulate blood loss in the research laboratory, participants will complete a test with their lower body in a custom-designed vacuum chamber for a brief period of time.

DETAILED DESCRIPTION:
Pain management on the battlefield is critical for the wellbeing of the soldier. Given that a hemorrhagic injury on the battlefield is virtually always associated with pain, it is paramount that the selected pain medication does not disrupt appropriate physiological mechanisms that are beneficial towards the maintenance of blood pressure and vital organ blood flow during that hemorrhagic insult. Current guidelines for the selection of pain medications of a hemorrhaging soldier are based upon limited scientific evidence, with the vast majority of supporting studies being conducted on anesthetized animals. Thus, the interaction between hemorrhagic shock and pain medications commonly employed on the battlefield is yet to be determined in the conscious humans.

This study will test the hypothesis that sufentanil will impair the capacity for a conscious human to tolerate a hemorrhagic insult.

The obtained data will provide the necessary scientific evidence in humans to support the Committee on Tactical Combat Casualty Care (CoTCCC) guidelines on the analgesic of choice for moderate to severe injuries where the casualty is in hemorrhagic shock. Notably, such data will identify the analgesic that least compromises a human's ability to tolerate a hemorrhagic insult, ultimately providing critical information to the combat medic on which analgesic should be employed for such an injury.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* Healthy
* Non-obese (body mass index less than 30 kg/m2)
* Body mass greater than or equal to 65 kg
* Speak English

Exclusion Criteria:

* Subjects not in the defined age range
* Subjects who have cardiac, respiratory, neurological and/or metabolic illnesses
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy or breast feeding
* Body mass less than 65 kg
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Subjects who cannot speak or read English
* Positive urine drug screen
* Currently taking pain modifying medication(s)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute for Exercise and Environmental Medicine, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Sufentanil: Participants received the placebo first followed by sufentanil.
- Sufentanil Then Placebo: Participants received the sufentanil first followed by placebo.
Period: Overall Study
Arm/Group | Placebo Then Sufentanil | Sufentanil Then Placebo
Started | 28 | 18
Completed | 20 | 9
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Participants in Crossover Design: Participants received both placebo and sufentanil in a randomized crossover model. Thus, the reported baseline characteristics reflect those individuals who participated in both limbs.
Arm/Group | Enrolled Participants in Crossover Design
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 2
  Unknown or Not Reported | 2
Body-Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25 (2)

OUTCOME MEASURES:

1. Primary Outcome: Tolerance to Simulated Hemorrhage
Description: Tolerance to a simulated hemorrhagic challenge will be assessed, for both the placebo and sufentanil limbs, by causing progressive central hypovolemia via lower-body negative pressure. This progressive lower-body negative pressure (LBNP) challenge will be performed until the onset of syncopal symptoms (defined as: profound bradycardia, a precipitous drop in arterial blood pressure and accompanying narrowing of pulse pressure, a sustained systolic blood pressure less than 80 mmHg, and/or subjective symptoms such as light-headedness, sweating, nausea, or dizziness). The primary variable will be the quantification of lower-body negative pressure that is required to cause these symptoms. This quantification will be objectively measured via a cumulative stress index which is calculated as the sum of the product of the LBNP level and the duration of each level, until test termination (i.e., 40 mmHg x 3 min + 50 mmHg x 3 min, etc).
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: min*mmHg
Arm/Group | Sufentanil | Placebo
Number analyzed (Participants) | 29 | 29
min*mmHg | 599 (412) | 651 (271)

2. Secondary Outcome: Pain Assessment
Description: Pain assessments will be conducted using a digital algometer to obtain maximum pain thresholds caused by pressure. This pain assessment technique is conducted by applying the tip of a hand-held digital algometer on the subject's digit. Force is gradually increased and the peak force is recorded when the subject first reports a painful sensation. Removal of the pressure from the algometer immediately relieves the painful sensation and the subject can voluntarily stop the test at any time. This assessment will be performed when the subject has received placebo and sufentanil.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sufentanil | Placebo
Number analyzed (Participants) | 29 | 29
kg | 1.04 (0.43) | 1.16 (0.40)

ADVERSE EVENTS:
Time Frame: Adverse data was collected over the 6 hours of the study.
Arm/Group | Sufentanil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04959812/Prot_SAP_002.pdf
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT04959812/ICF_001.pdf